CLINICAL TRIAL: NCT03188185
Title: A Phase 3b Efficacy and Safety Study of Adjunctive ALKS 5461 in Treatment Refractory Major Depressive Disorder
Brief Title: A Study of ALKS 5461 for Treatment Refractory Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK5461-217
Record Dates: First submitted 2017-06-09; First posted 2017-06-15 (Actual); Results first posted 2021-03-15 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Major Depressive Disorder
Keywords: Alkermes; Major Depressive Disorder; Treatment Refractory MDD; ALKS 5461
MeSH Terms: conditions — Depressive Disorder, Major | interventions — ALKS 5461

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALKS 5461 (Experimental): Sublingual tablets
  Interventions: Drug: ALKS 5461
- ALKS 5461 Placebo (Placebo Comparator): Sublingual tablets
  Interventions: Drug: ALKS 5461 Placebo

INTERVENTIONS:
Drug: ALKS 5461 — Samidorphan + buprenorphine, administered sublingually
  Arms: ALKS 5461
Drug: ALKS 5461 Placebo — Placebo tablet, administered sublingually
  Arms: ALKS 5461 Placebo

SUMMARY:
This study will evaluate the efficacy, safety, and tolerability of adjunctive ALKS 5461 in adults who have treatment refractory MDD.

ELIGIBILITY:
Inclusion Criteria:

* Have a Major Depressive Disorder (MDD) primary diagnosis
* Have a body mass index (BMI) of 18.0 to </= 40.0 kg/m^2
* Be willing and able to follow the study procedures and visits as outlined in the protocol (including agreeing not to enroll in any other clinical trials)
* Have inadequate responses to antidepressant therapy (ADT) in the current Major Depressive Episode (MDE)
* Additional criteria may apply

Exclusion Criteria:

* Has any finding that would compromise the safety of the subject or affect their ability to adhere to the protocol visit schedule or fulfill visit requirements
* Has any other significant medical condition (eg, neurological, psychiatric, or metabolic) or clinical symptom that could unduly risk the subject or affect the interpretation of study data
* Has any current primary diagnosis other than MDD, where primary diagnosis is defined as the primary source of current distress and functional impairment
* Has experienced hallucinations, delusions, or any psychotic symptoms in the current MDE
* Has been hospitalized for MDD within 3 months before screening
* Has used opioid agonists (eg, codeine, oxycodone, tramadol, morphine) or opioid antagonists (eg, naloxone, naltrexone) within 14 days prior to screening
* Has received electroconvulsive therapy treatment within the last 2 years or within the current MDE or failed a course of electroconvulsive treatment at any time
* Has a significant risk for suicide
* Has a positive breath alcohol test at screening
* Has a positive test for drugs of abuse at screening or visit 2
* Is pregnant, planning to become pregnant, or is breastfeeding during the study
* Additional criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Pathak, MD, Study Director — Alkermes, Inc.
Locations (34):
- United States (30):
  - Alkermes Investigational Site, Tucson, Arizona
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Los Alamitos, California
  - Alkermes Investigational Site, Oceanside, California
  - Alkermes Investigational Site, Pico Rivera, California
  - Alkermes Investigational Site, Redlands, California
  - Alkermes Investigational Site, Santa Ana, California
  - Alkermes Investigational Site, Sherman Oaks, California
  - Alkermes Investigational Site, Temecula, California
  - Alkermes Investigative Site, Upland, California
  - Alkermes Investigational Site, Hollywood, Florida
  - Alkermes Investigational Site, Jacksonville, Florida
  - Alkermes Investigational Site, Lauderhill, Florida
  - Alkermes Investigational Site, Orlando, Florida
  - Alkermes Investigative Site, Palm Bay, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Decatur, Georgia
  - Alkermes Investigational Site, Pikesville, Maryland
  - Alkermes Investigational Site, O'Fallon, Missouri
  - Alkermes Investigational Site, Jamaica, New York
  - Alkermes Investigational Site, Mount Kisco, New York
  - Alkermes Investigational Site, Canton, Ohio
  - Alkermes Investigational Site, Cincinnati, Ohio
  - Alkermes Investigational Site, Oklahoma City, Oklahoma
  - Alkermes Investigational Site, Allentown, Pennsylvania
  - Alkermes Investigational Site, Memphis, Tennessee
  - Alkermes Investigational Site, Dallas, Texas
  - Alkermes Investigational Site, DeSoto, Texas
  - Alkermes Investigational Site, Woodstock, Vermont
  - Alkermes Investigative Site, Bellevue, Washington
- Australia (3):
  - Alkermes Investigational Site, Frankston, Victoria
  - Alkermes Investigational Site, Noble Park, Victoria
  - Alkermes Investigational Site, Richmond, Victoria
- Alkermes Investigational Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were diagnosed with treatment refractory major depressive disorder (MDD), defined as having at least 2 inadequate responses to commercially available antidepressant therapies (ADTs) during the current major depressive episode (MDE). All subjects continued to take an approved ADT for the duration of the study.
Pre-assignment Details: This was a Sequential Parallel Comparison Design (SPCD) study comprised of 2 stages. In Stage 1 subjects were randomized to ALKS 5461 or placebo. In Stage 2 only placebo non-responders from Stage 1 were re-randomized to ALKS 5461 or placebo.
Groups:
- S1: Placebo: Randomized to placebo in Stage 1
- S1: ALKS 5461 2mg/2mg: Randomized to ALKS 5461 2mg/2mg in Stage 1
- S2: Placebo: Randomized to placebo in Stage 2
- S2: ALKS 5461 2mg/2mg: Randomized to ALKS 5461 2mg/2mg in Stage 2
Period: Stage 1
Arm/Group | S1: Placebo | S1: ALKS 5461 2mg/2mg | S2: Placebo | S2: ALKS 5461 2mg/2mg
Started | 198 | 80 | 0 | 0
Completed | 179 | 64 | 0 | 0
Not Completed | 19 | 16 | 0 | 0
Not completed — Adverse Event | 4 | 12 | 0 | 0
Not completed — Lack of Efficacy | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 6 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0 | 0
Not completed — Identified as a professional patient | 0 | 1 | 0 | 0
Period: Stage 2
Arm/Group | S1: Placebo | S1: ALKS 5461 2mg/2mg | S2: Placebo | S2: ALKS 5461 2mg/2mg
Started | 0 | 0 | 64 | 63
Completed | 0 | 0 | 55 | 57
Not Completed | 0 | 0 | 9 | 6
Not completed — Adverse Event | 0 | 0 | 2 | 4
Not completed — Lack of Efficacy | 0 | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | S1: Placebo | S1: ALKS 5461 2mg/2mg | Total
Number analyzed (Participants) | 198 | 80 | 278
Age, Continuous [Median (Full Range); unit: years] | 44 [18 to 67] | 40.5 [18 to 70] | 43 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 57 | 196
  Male | 59 | 23 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 10 | 41
  Not Hispanic or Latino | 167 | 70 | 237
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 9 | 33
  White | 160 | 63 | 223
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 5 | 2 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 176 | 72 | 248
  Australia | 22 | 8 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the End of Treatment (EOT) in the Montgomery Asberg Depression Rating Scale-10 (MADRS-10) Scores
Description: The MADRS-10 scale is a clinician-administered questionnaire comprised of 10 items used to measure the severity of Major Depressive Disorder (MDD) symptoms. Scores range from 0 (no apparent symptoms) to 60 (most severe symptoms). Individual questionnaire items include: Apparent Sadness, Reported Sadness, Inner Tension, Reduced Sleep, Reduced Appetite, Concentration Difficulties, Lassitude, Inability to Feel, Pessimistic Thoughts, and Suicidal Thoughts.
Time Frame: Baseline and 5 weeks for Stage 1, Baseline and 6 weeks for Stage 2
Population: Stage 1 and Stage 2 Full Analysis Sets (FAS) consisted of subjects who were randomized and took at least 1 dose of study drug and had at least 1 postbaseline MADRS assessment in the respective stage.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | S1: Placebo | S1: ALKS 5461 2mg/2mg | S2: Placebo | S2: ALKS 5461 2mg/2mg
Number analyzed (Participants) | 195 | 76 | 64 | 63
score on a scale | -11.4 (0.70) | -13.9 (1.12) | -4.2 (1.06) | -4.7 (1.11)
Statistical Analysis 1: Comparison: S1: Placebo vs S1: ALKS 5461 2mg/2mg vs S2: Placebo vs S2: ALKS 5461 2mg/2mg; Analysis was conducted for each stage separately, and overall efficacy was based on combined stage analysis where stage-specific estimates were combined using pre-specified equal weights. Within each stage ALKS 5461 2mg/2mg was compared to placebo (i.e., ALKS 5461 2mg/2mg S1 vs Placebo S1; and ALKS 5461 2mg/2mg S2 vs Placebo S2); Test type: Superiority — Hypothesis tests were two-sided with an alpha of 0.05; p = 0.128, Mixed Models Analysis — ALK 5461 was compared to placebo using stage-specific MMRM for MADRS-10 Change from Baseline.Model-derived estimates were combined using equal weights; Least Squares Mean Difference = -1.5, 95% CI 2-sided [-3.5 to 0.4], Standard Error of Mean 0.99

2. Secondary Outcome: Montgomery Asberg Depression Rating Scale (MADRS) Response Rate
Description: The percentage of subjects demonstrating a MADRS-10 treatment response, defined as a >/= 50% reduction in MADRS-10 score from baseline to the end of the efficacy period (Week 5 for Stage 1, Week 6 for Stage 2). The MADRS-10 scale is a measure of the severity of Major Depressive Disorder (MDD) symptoms and includes the following 10 items: Apparent Sadness, Reported Sadness, Inner Tension, Reduced Sleep, Reduced Appetite, Concentration Difficulties, Lassitude, Inability to Feel, Pessimistic Thoughts, and Suicidal Thoughts. Scores range from 0 (no apparent symptoms) to 60 (most severe symptoms).
Time Frame: Baseline and 5 weeks for Stage 1, Baseline and 6 weeks for Stage 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | S1: Placebo | S1: ALKS 5461 2mg/2mg | S2: Placebo | S2: ALKS 5461 2mg/2mg
Number analyzed (Participants) | 195 | 76 | 64 | 63
Participants
  Yes | 53 | 27 | 10 | 11
  No | 142 | 49 | 54 | 52

3. Secondary Outcome: Montgomery Asberg Depression Rating Scale (MADRS) Remission Rate
Description: The percentage of subjects achieving remission, defined as a subject with a score </= 10 at the end of the efficacy period (Week 5 for Stage 1, Week 6 for Stage 2). The MADRS-10 scale is a measure of the severity of Major Depressive Disorder (MDD) symptoms and includes the following 10 items: Apparent Sadness, Reported Sadness, Inner Tension, Reduced Sleep, Reduced Appetite, Concentration Difficulties, Lassitude, Inability to Feel, Pessimistic Thoughts, and Suicidal Thoughts. Scores range from 0 (no apparent symptoms) to 60 (most severe symptoms).the end of the efficacy period.
Time Frame: 5 weeks for Stage 1, 6 weeks for Stage 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | S1: Placebo | S1: ALKS 5461 2mg/2mg | S2: Placebo | S2: ALKS 5461 2mg/2mg
Number analyzed (Participants) | 195 | 76 | 64 | 63
Participants
  Yes | 31 | 14 | 10 | 8
  No | 164 | 62 | 54 | 55

ADVERSE EVENTS:
Time Frame: 5 weeks for Stage 1 and 6 weeks for Stage 2
Description: The safety population includes all subjects who were randomized and received at least 1 dose of study drug.
Arm/Group | S1: Placebo | S1: ALKS 5461 2mg/2mg | S2: Placebo | S2: ALKS 5461 2mg/2mg
All-Cause Mortality (participants affected / at risk) | 0/198 | 0/80 | 0/64 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/198 | 1/80 | 1/64 | 0/63
Other Adverse Events (participants affected / at risk) | 43/198 | 56/80 | 3/64 | 29/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | S1: Placebo (N=198) | S1: ALKS 5461 2mg/2mg (N=80) | S2: Placebo (N=64) | S2: ALKS 5461 2mg/2mg (N=63)
Serotonin Syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | S1: Placebo (N=198) | S1: ALKS 5461 2mg/2mg (N=80) | S2: Placebo (N=64) | S2: ALKS 5461 2mg/2mg (N=63)
Nausea (Gastrointestinal disorders) | 10 | 29 | 0 | 16
Constipation (Gastrointestinal disorders) | 2 | 9 | 0 | 3
Vomiting (Gastrointestinal disorders) | 4 | 5 | 0 | 6
Dizziness (Nervous system disorders) | 4 | 18 | 0 | 8
Somnolence (Nervous system disorders) | 5 | 10 | 1 | 3
Headache (Nervous system disorders) | 14 | 9 | 0 | 7
Sedation (Nervous system disorders) | 5 | 8 | 0 | 3
Abnormal dreams (Psychiatric disorders) | 3 | 4 | 0 | 3
Fatigue (General disorders) | 3 | 4 | 1 | 2
Nasopharyngitis (Infections and infestations) | 5 | 4 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT03188185/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT03188185/SAP_001.pdf